CLINICAL TRIAL: NCT02603237
Title: Metabolic Response to Fat and Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Rima Obeid, Prof. (apl.) Dr., Universität des Saarlandes
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Postprandial metabolomics
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Insulin Resistance; Healthy
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose tolerance test (Other): All participants will receive an oral standardized glucose tolerance test
  Interventions: Other: Glucose tolerance test
- Fat tolerance test (Other): The same participants will receive an oral standardized fat load test
  Interventions: Other: Fat tolerance test

INTERVENTIONS:
Other: Glucose tolerance test — Standardized oral glucose tolerance test (75 g oral glucose) and blood collection before and 2hrs after the glucose load
  Arms: Glucose tolerance test
Other: Fat tolerance test — Oral fat tolerance will be provided to fasting participants and blood samples will be collected before and 4 hrs after the fat load.
  Arms: Fat tolerance test

SUMMARY:
The study will compare plasma and urine post-prandial metabolomics after fat and glucose oral load according to lifestyle factors.

DETAILED DESCRIPTION:
The metabolic response in plasma and urine, pre- and post-load tests in people with specific dietary lifestyles will be tested. This project will focus on fat and glucose induced changes of targeted metabolic pathways that have been related to diabetes and obesity risk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* On a stable dietary habits

Exclusion Criteria:

* Pregnancy
* Malabsorption disorders
* Present or former cancer
* Any oral medication that affect glucose or fat absorptions
* Cholesterol lowering drugs (i.e. Statins)
* other drugs: fibrates, MTX, or vitamin supplements
* Diabetes (type 1 and type 2)
* Alcoholism
* Weight losing diet during the last 4 months
* Liver diseases
* Renal dysfunction
* Gastric resection.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Plasma levels of branched chain amino acid | Changes between baseline and 2 hours
Plasma Trimethylamin N-oxide | Changes between baseline and 2 hours
Plasma glucose level | Changes between baseline and 2 hours
Plasma glucose | Changes between baseline and 2 hours
Plasma level of acetyl-CoA | Changes between baseline and 2 hours

SECONDARY OUTCOMES:
Plasma malonyl-CoA | Changes between baseline and 2 hours
Plasma phosphatidylcholine | Changes between baseline and 2 hours
Plasma insulin | Changes between baseline and 2 hours
Plasma leptin | Changes between baseline and 2 hours
Plasma Lactate | Changes between baseline and 2 hours
Plasma pyruvate | Changes between baseline and 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rima Obeid, Study Director — Universität des Saarlandes
Locations (1):
- University of Saarland, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Undecided
will be decided at a later stage